CLINICAL TRIAL: NCT06958991
Title: Confocal Histolog Scanner in Routine Breast-Conserving Surgery
Brief Title: Confocal Histolog Scanner in Routine Breast-Conserving Surgery (CHiB)
Acronym: CHiB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Fribourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-D0101; 20240829 (Other Grant/Funding Number: SamanTree)
Record Dates: First submitted 2025-04-13; First posted 2025-05-06 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Invasive; Breast Cancer Surgery; Lumpectomy; Confocal Laser Endomicroscopy
Keywords: breast cancer surgery; confocal microscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast Cancer patient with Lumpectomy (Experimental): The clinical performance study is collecting data from the use of a CE mark product used within the scope of its intended purpose to intraoperatively visualize tissue specimen. The subjects are not submitted to invasive and burdensome procedures compared to the standard of care surgical practices and regular use of the CE mark product.
  Interventions: Device: Histolog Scanner

INTERVENTIONS:
Device: Histolog Scanner — The clinical performance study is collecting data from the use of a CE mark product used within the scope of its intended purpose to intraoperatively visualize tissue specimen. The subjects are not submitted to invasive and burdensome procedures compared to the standard of care surgical practices and regular use of the CE mark product.

SUMMARY:
The clinical performance study is collecting data from the use of a CE mark product used within the scope of its intended purpose to intraoperatively visualize tissue specimen. The subjects are not submitted to invasive and burdensome procedures compared to the standard of care surgical practices and regular use of the CE mark product.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. Moreover, numerous women have the diagnosis of a ductal carcinoma in situ (DCIS) each year, which can develop to invasive breast cancer without therapy. Breast conserving surgery (BCS) is the most performed surgical treatment for women with early-stage breast cancer and/ or DCIS. There is an ongoing need for more immediate and accurate methods for the intraoperative assessment (IOA) of breast tissue margins to achieve tumor free margins. A method for rapidly and accurately identifying positive surgical margins intraoperatively would allow the surgeon to immediately excise additional tissue to achieve negative margins. Thereby sparing the Subject a reoperation with all following consequences i.e., reduced oncological safety, reduced cosmetic, and economic burden. The Histolog® Scanner (HLS), a confocal laser scanning microscope was developed with the CE Mark intended use of imaging excised human tissue specimens to visualize morphological microstructures. Such a feature allows real-time IOA offering cutting edge imaging support beyond the conventional imaging techniques in clinical decision making. Promising results have been previously obtained in the SENOSI study of Sion (Switzerland) and the POLARHIS and HELIXIR studies in Germany. Therefore, this study is proposed to evaluate in real life the reoperation rates (ROR) of breast cancer and/or DCIS surgery when the HLS is used in the context of breast tissue margin assessment.

Primary Objective:

Evaluate the proportion of patients that had a surgical reoperation due to cancer-positive margins (Reoperation Rate).

Secondary Objectives:

Detection Rate

* To evaluate real life detection of breast cancerwhen the HLS and accessories are used intraoperatively by surgeons for the assessment of breast surgical specimens in comparison with the final pathology assessment (gold standard) Usability
* To survey usability of the HLS and accessories when used intraoperatively by surgeons for the assessment of breast surgical specimens Economic Impact
* To evaluate the economic impact for the hospitals/payers of the reoperation rate achieved by the use of the HLS and accessories for the assessment of breast surgical specimens Safety
* To monitor the safety of HLS and accessories when used intraoperatively by surgeons for the assessment of breast surgical specimens

Primary Endpoint:

Reoperation Rate

- Proportion of women who had a reoperation because of cancer positive margins identified at final pathology assessment.

Secondary Endpoints:

Detection Rate

* Proportion of women for whom an unsafe margin was detected with HLS
* Agreement between margin cancerous status of the main surgical specimen and of recuts determined intraoperatively with the HLS and postoperative final pathology assessment using histological slides
* Rates of the intraoperative recuts depending on the different evaluation tools (HLS, ultrasound and specimen radiography)
* Weight and dimensions of surgical specimens
* HLS usage time on surgical specimens and recuts Usability
* Usability rates of HLS and accessories including image acquisition, processing, and analysing time
* Relevant tissue microstructures recognition by surgeons/ user
* HLS and accessories ease of use
* Rate of HLS' damage to tissue specimens

Economic Impact

- Change in hospital cost per patient with BCS with or without using the HLS and accessories. This will be evaluated by monitoring the costs of breast conserving surgeries and the costs related to the use of the HLS including device price, HLS consumables, time of use of the HLS, reoperation rates and their associated surgical resources.

Safety

- Incidence of adverse device effects during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult female Subject ≥18 years old.
* Subject scheduled for breast conserving surgery of invasive and/or in-situ ductal and lobular carcinoma.
* Subject is able to read, understand and sign the informed consent.

Exclusion Criteria:

* Subject with planned mastectomy
* Subject does not speak French- Subject with planned tumor-adapted breast reduction
* Subject is pregnant/ lactating. Subjects pregnant/lactating are excluded because such subjects are presenting additional risks during the surgery and they are also rare.
* Participation in any other clinical study that would affect data acquisition.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Sex and gender are not a relevant variable in this study because it focuses exclusively on cisgender women with BCS.
Enrollment: 100 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Reoperation Rate | From enrollment to the end of treatment (surgery) at 1 month
  Proportion of women who had a reoperation because of cancer positive margins identified at final pathology assessment.

SECONDARY OUTCOMES:
Detection Rate | 1 year
  - Agreement between margin cancerous status of the main surgical specimen and of recuts determined intraoperatively with the HLS and postoperative final pathology assessment using histological slides (sensibility and specificity)
Usability | 1 year
  - Usability rates of HLS and accessories: analysis time
Economic Impact | 1 year
  - Change in hospital cost per patient with BCS with or without using the HLS and accessories. This will be evaluated by comparing the usual average cost of breast conserving surgeries and the costs related to the use of the HLS during the surgery
Incidence of adverse device effects | 14 month
  Incidence of adverse device effects during the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- HFR, Villars-sûr-glâne, Canton of Fribourg, Switzerland